CLINICAL TRIAL: NCT06608290
Title: Association Between the Application of Parasternal Blockade and Serum Lactate Level in Trans and Post-anesthetic Stages in Cardiac Surgery.
Brief Title: Paraesternal Blockade and Lactate Serum Levels in Patients with Cardiac Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Clotilde Fuentes-Orozco, Investigador Principal, Instituto Mexicano del Seguro Social
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2023-1301-024.
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2023-09

CONDITIONS: Parasternal Block; Cardiac Surgery; Serum Lactate
Keywords: Parasternal block; cardiac surgery; serum lactate; cardiopulmonary bypass; cardiovascular surgery post-surgical unit

STUDY DESIGN:
Intervention Model Description: Patients were classified as a group of cases with parasternal blockade and as a group of controls without parasternal blockade, with a ratio of cases to controls of 1:1. In the case-control groups, patients with elevated serum lactate levels greater than 2 mmol/L and those who remained below this limit were identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blockade (Experimental): In patients which parasternal block has been applied
  Interventions: Procedure: parasternal block; Diagnostic Test: Lactate serum level
- Control (Experimental): In patients which parasternal block has not been applied
  Interventions: Diagnostic Test: Lactate serum level

INTERVENTIONS:
Procedure: parasternal block — Administration of parasternal block with ropivacaine, bilaterally at the sternum before the start of surgery.
  Arms: Blockade
Diagnostic Test: Lactate serum level — Blood samples were taken to identify serum lactate levels greater than 2 mmol/l and those that remained below this limit.

SUMMARY:
Parasternal blockade has been related to a reduction of the postoperative inflammatory response, by inhibition of the stress response, leading to a better prognosis. Increased lactate level is a useful parameter in identifying patients at risk of postoperative morbidity and mortality. The objective was to evaluate the association between parasternal blockade and serum lactate level in patients undergoing cardiac surgery, both trans- and post-anesthesia. 86 patients between 60-70 years of age participated. An association was found between the application of parasternal blockade in cardiac surgery and the presence of lower trans and postanesthetic serum lactate levels.

DETAILED DESCRIPTION:
An analytical cross-sectional study in adult patients who underwent elective cardiac surgery. A total sample of 86 patients was obtained, 43 in the case group and 43 in the control group. Adult patients older than 18 years, of either sex, with ASA II-III, patients who underwent cardiac surgery with median sternotomy and use of cardiopulmonary bypass were included.

ELIGIBILITY:
Inclusion criteria

* Adult patients over 18 years of age
* Either sex
* ASA II-IV
* Patients who underwent cardiac surgery with median sternotomy and use of cardiopulmonary bypass.

Elimination criteria

- Patients with pre-existing conditions that could independently affect serum lactate levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Lactate serum levels | 24 Hours
  Blood samples were taken to identify serum lactate levels greater than 2 mmol/l and those that remained below this limit.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación Biomédica 02, Unidad Médica de alta especialidad, Hospital de Especialidades Centro Médico Nacional de Occidente, Instituto Mexicano del Seguro Social, Guadalajara 44329, México, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
This is a closed study completed at a single center.

REFERENCES:
- [Background] Seghrouchni A, Atmani N, Moutakiallah Y, Belmekki A, El Bekkali Y, Houssa MA. Does severe hyperlactatemia during cardiopulmonary bypass predict a worse outcome? Ann Med Surg (Lond). 2021 Dec 21;73:103198. doi: 10.1016/j.amsu.2021.103198. eCollection 2022 Jan. PMID 35070281
- [Background] Zhou Y, Yang C, Jin Z, Zhang B. Intraoperative use of cell saver devices decreases the rate of hyperlactatemia in patients undergoing cardiac surgery. Heliyon. 2023 May 4;9(5):e15999. doi: 10.1016/j.heliyon.2023.e15999. eCollection 2023 May. PMID 37215823
- [Background] Yang HH, Chang JC, Jhan JY, Cheng YT, Huang YT, Chang BS, Chao SF. Prognostic value of peak lactate during cardiopulmonary bypass in adult cardiac surgeries: A retrospective cohort study. Tzu Chi Med J. 2020 Feb 27;32(4):386-391. doi: 10.4103/tcmj.tcmj_215_19. eCollection 2020 Oct-Dec. PMID 33163386
- [Background] Wang D, Wang S, Wu J, Le S, Xie F, Li X, Wang H, Huang X, Du X, Zhang A. Nomogram Models to Predict Postoperative Hyperlactatemia in Patients Undergoing Elective Cardiac Surgery. Front Med (Lausanne). 2021 Dec 2;8:763931. doi: 10.3389/fmed.2021.763931. eCollection 2021. PMID 34926506
- [Background] Li JQ, Li ZH, Dong P, Liu P, Xu YZ, Fan ZJ. Effects of parasternal intercostal block on surgical site wound infection and pain in patients undergoing cardiac surgery: A meta-analysis. Int Wound J. 2023 Oct 17;21(2):e14433. doi: 10.1111/iwj.14433. Online ahead of print. PMID 37846438
- [Background] Wong HMK, Chen PY, Tang GCC, Chiu SLC, Mok LYH, Au SSW, Wong RHL. Deep Parasternal Intercostal Plane Block for Intraoperative Pain Control in Cardiac Surgical Patients for Sternotomy: A Prospective Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2024 Mar;38(3):683-690. doi: 10.1053/j.jvca.2023.11.038. Epub 2023 Nov 30. PMID 38148266
- [Background] Chen Y, Li Q, Liao Y, Wang X, Zhan MY, Li YY, Liu GJ, Xiao L. Preemptive deep parasternal intercostal plane block for perioperative analgesia in coronary artery bypass grafting with sternotomy: a randomized, observer-blind, controlled study. Ann Med. 2023;55(2):2302983. doi: 10.1080/07853890.2024.2302983. Epub 2024 Feb 20. PMID 38375661
- [Background] Bhat HA, Khan T, Puri A, Narula J, Mir AH, Wani SQ, Ashraf HZ, Sidiq S, Kabir S. To evaluate the analgesic effectiveness of bilateral erector spinae plane block versus thoracic epidural analgesia in open cardiac surgeries approached through midline sternotomy. J Anesth Analg Crit Care. 2024 Mar 1;4(1):17. doi: 10.1186/s44158-024-00148-4. PMID 38429852
- [Background] Caruso TJ, Lawrence K, Tsui BCH. Regional anesthesia for cardiac surgery. Curr Opin Anaesthesiol. 2019 Oct;32(5):674-682. doi: 10.1097/ACO.0000000000000769. PMID 31356362
- [Background] Miao Q, Wu DJ, Chen X, Xu M, Sun L, Guo Z, He B, Wu J. Target blood pressure management during cardiopulmonary bypass improves lactate levels after cardiac surgery: a randomized controlled trial. BMC Anesthesiol. 2021 Dec 8;21(1):309. doi: 10.1186/s12871-021-01537-w. PMID 34879822
- [Background] Padala SRAN, Badhe AS, Parida S, Jha AK. Comparison of preincisional and postincisional parasternal intercostal block on postoperative pain in cardiac surgery. J Card Surg. 2020 Jul;35(7):1525-1530. doi: 10.1111/jocs.14651. Epub 2020 Jun 24. PMID 32579779
- [Background] Schiavoni L, Nenna A, Cardetta F, Pascarella G, Costa F, Chello M, Agro FE, Mattei A. Parasternal Intercostal Nerve Blocks in Patients Undergoing Cardiac Surgery: Evidence Update and Technical Considerations. J Cardiothorac Vasc Anesth. 2022 Nov;36(11):4173-4182. doi: 10.1053/j.jvca.2022.07.025. Epub 2022 Jul 24. PMID 35995636
- [Background] Abadi A, Cohen R. Evaluation of an Enhanced Recovery After Surgery Protocol Including Parasternal Intercostal Nerve Block in Cardiac Surgery Requiring Sternotomy. Am Surg. 2021 Dec;87(10):1561-1564. doi: 10.1177/00031348211024638. Epub 2021 Jun 23. PMID 34162242
- [Background] Demir AZ, Ozgok A, Balci E, Karaca OG, Simsek E, Gunaydin S. Preoperative ultrasound-guided bilateral thoracic erector spinae plane block within an enhanced recovery program is associated with decreased intraoperative lactate levels in cardiac surgery. Perfusion. 2024 Mar;39(2):324-333. doi: 10.1177/02676591221140754. Epub 2022 Nov 21. PMID 36408617
- [Background] Bloc S, Perot BP, Gibert H, Law Koune JD, Burg Y, Leclerc D, Vuitton AS, De La Jonquiere C, Luka M, Waldmann T, Vistarini N, Aubert S, Menager MM, Merzoug M, Naudin C, Squara P. Efficacy of parasternal block to decrease intraoperative opioid use in coronary artery bypass surgery via sternotomy: a randomized controlled trial. Reg Anesth Pain Med. 2021 Aug;46(8):671-678. doi: 10.1136/rapm-2020-102207. Epub 2021 May 14. PMID 33990437
- [Background] Liu H, Emelife PI, Prabhakar A, Moll V, Kendrick JB, Parr AT, Hyatali F, Pankaj T, Li J, Cornett EM, Urman RD, Fox CJ, Kaye AD. Regional anesthesia considerations for cardiac surgery. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):387-406. doi: 10.1016/j.bpa.2019.07.008. Epub 2019 Jul 17. PMID 31791558